CLINICAL TRIAL: NCT01248026
Title: Impact of Buttermilk on Cholesterol Concentration and Homeostasis
Acronym: BMILK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Dairy Farmers of Canada (Other)
Responsible Party: Principal Investigator, Benoit Lamarche, Professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INAF-2010-035
Record Dates: First submitted 2010-11-18; First posted 2010-11-25 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular disease; Buttermilk; Blood lipids; Cholesterol absorption; Cholesterol synthesis
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Buttermilk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buttermilk (Experimental)
  Interventions: Other: Buttermilk
- Placebo (Placebo Comparator)
  Interventions: Other: Buttermilk

INTERVENTIONS:
Other: Buttermilk — Consumption of the 2 experimental periods
  1. buttermilk (45 g/d)
  2. placebo (45 g/d,)
  Other Names: chocolat buttermilk ready-to-use pouches

SUMMARY:
The role of low-density lipoprotein cholesterol (LDL-C) in the pathogenesis of cardiovascular disease (CVD) and the clinical benefit of lowering LDL-C in high-risk patients have both been well established. The key contribution of the intestine to whole body cholesterol homeostasis and thus to regulating plasma cholesterol concentrations has also been recognized over the last years. It is now clear that cholesterol homeostasis and hence plasma LDL-C concentrations are maintained by a fine-tuned balance between intestinal cholesterol absorption and endogenous cholesterol synthesis.

Cholesterol is a highly hydrophobic molecule and for that reason, its absorption is almost entirely dependent on its solubilizing capacity in bile acid micelles within the intestine. Recent in vitro studies from our laboratory have shown that buttermilk, a unique by-product of butter manufacturing resulting from the churning of cream, has a strong inhibitory effect on cholesterol micelle solubility. This phenomenon is likely due to the presence of unique milk fat globule membrane (MFGM) fragments present in buttermilk that are produced during the manufacturing of dairy cream into butter. Most of the work done so far on the subject has focused on phospholipids purified from MFGM, while overlooking the complex and entire MFGM mixture of bioactive proteins and polar lipids found in buttermilk. To the best of our knowledge, no study has yet documented the impact of whole buttermilk on plasma cholesterol concentration in human.

The general objective of this research project is to investigate for the first time the impact of buttermilk on plasma cholesterol and other risk factors for CVD in humans. More specifically, we propose to investigate the impact of buttermilk consumption on plasma LDL-C and other CVD risk factors as well as on plasma surrogates of cholesterol absorption and synthesis.

DETAILED DESCRIPTION:
The proposed research will be undertaken as a double-blind randomized cross-over study with participants being subjected to 2 consecutive treatments of 4 weeks each, in random order, during which they will consume 45g of buttermilk and a macro- and micronutrient matching placebo. The treatments will be different in their content of MFGM (present in buttermilk, absent in placebo). Buttermilk and placebo will be fully characterized and formulated in ready-to-use pouches, each pouch containing 22.5 g of artificially flavored products that will have to be mixed in a fixed amount of water for consumption. Participants will have to consume two pouches every day. Based on a 2500 kcal/day regimen, we have calculated that these placebo and buttermilk formulation will contribute to approximately 200 kcal (from 5% and 10%) of the daily energy intake of participants, who will be asked to maintain other aspects of their nutritional habits constant throughout the study.

Fluctuations in female hormones have been shown to influence metabolic variables. For that reason, outcomes at the end of each dietary phase will be measured during the follicular phase of menstrual cycle (day 3 to day 9) in pre-menopausal women. This is another argument for using a 4-wk intervention, which essentially corresponds to the mean duration of the menstrual cycle of most women. Pre-menopausal women will start the first diet during the first week of their menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged between 18 and 65 years
* For pre-menopausal women: regular menstrual cycle for the last 3 months (25- 35 days), using or not contraceptive agents
* LDL-Cholesterol concentration between 3.2 and 4.5 mmol/L
* A 10-yr calculated Framingham risk below 10%.
* Stable body weight (+/- 2 kg) for 6 months before the beginning of the study
* Smoking or not

Exclusion Criteria:

* Previous history of cardiovascular disease, type 2 diabetes and monogenic dyslipidemia
* Subjects taking medications for hyperlipidemia or hypertension
* Endocrine disorders
* Body mass index > 35 kg/m2
* Food allergies
* Men and women with extreme nutritional habits such as vegetarism or alcohol consumption > 2 drinks/day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in plasma LDL-Cholesterol concentrations | At the beginning of the study and the end of the 2 four-week periods

SECONDARY OUTCOMES:
Change in blood lipids (Total cholesterol, HDL-Cholesterol, Triglycerides) | At the beginning of the study and the end of the 2 four-week periods
Change in blood pressure | At the beginning of the study and the end of the 2 four-week periods
Change in surrogates of cholesterol absorption and synthesis | At the beginning of the study and the end of the 2 four-week periods
Change in anthropometric measures (waist and hip circumferences) | At the beginning of the study and the end of the 2 four-week periods

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD, FRCP (C, PhD), Study Director — Faculty of Medicine, Laval University
Locations (1):
- Institute of Nutraceutical and Functional Foods (INAF), Laval University, Québec, Quebec, Canada

REFERENCES:
- [Derived] Conway V, Couture P, Richard C, Gauthier SF, Pouliot Y, Lamarche B. Impact of buttermilk consumption on plasma lipids and surrogate markers of cholesterol homeostasis in men and women. Nutr Metab Cardiovasc Dis. 2013 Dec;23(12):1255-62. doi: 10.1016/j.numecd.2013.03.003. Epub 2013 Jun 17. PMID 23786821